CLINICAL TRIAL: NCT06831227
Title: Effect of High-Power Laser Therapy on the Size of Herniated Disc and Functional Outcome in Patients with Lumbosacral Radiculopathy.
Brief Title: High Power Laser Therapy for Herniated Disc and Lumbosacral Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, wessam abelfattah mohamed alrefaie, assistant lecture of Physical Therapy for Neurology and Neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pٌٌ.T.REC/012/005509
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Herniated Lumbar Disc
Keywords: High Power Laser; Herniated disc; LUMBOSACRAL RADICULOPATHY
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPLT (Active Comparator): this group will receive high power laser therapy (HPLT) for 20 minutes in addition to selected physical therapy exercise program 25 minutes and hot pack ten for 18 sessions three times weekly for 6 weeks.
  Interventions: Device: High power Laser Therapy; Device: physical therapy exercise program and hot pack
- physical therapy exercise program and hot pack (Sham Comparator): This group will receive the same selected physical therapy exercise program (45 minutes) and hot pack (10 min) for 18 session. All patients will attend the physical therapy clinic three times weekly for 6 weeks
  Interventions: Device: physical therapy exercise program and hot pack

INTERVENTIONS:
Device: High power Laser Therapy — A total course protocol: 18 sessions, for 6 weeks ,3 sessions per week. Patients will receive High power Laser treatment. manually set to bio stimulation mode with high peak power (5 - 6 W), energy per impulse 150 mJ/c2, wavelength measuring 1064 nm, and spot beam diameter area of 1 cm2.
  The hand piece was positioned in contact with and perpendicular to the treated area with the patient inside lying position with knee to chest. Scanning will perform transversely and longitudinally paravertebral region on the lower lumbar area at the level of the disc concerned. Each session included three phases (fast scan, sensitive trigger points, slow scan) and had a total duration of 20 minutes. During each session, a total energy of 3000 J was applied through three phases of treatment.
  Arms: HPLT
Device: physical therapy exercise program and hot pack — this group will receive the same selected physical therapy exercise program (45 minutes) and hot pack (10 min) for 18 session. All patients will attend the physical therapy clinic three times weekly for 6 weeks

SUMMARY:
To determine the effect of high-power laser therapy on the size of herniated disc and functional outcome in patients with lumbosacral radiculopathy.

DETAILED DESCRIPTION:
A herniated disc is a condition in which annulus fibrosus is damaged enabling the nucleus pulposus (which is normally located within the center of the disc) to herniate. It is a common cause of back pain. Unlike mechanical back pain, herniated disc pain is often burning or stinging, and may radiate into the lower extremity. Furthermore, in more severe cases, there can be associated with weakness or sensation changes. herniated disc injury may compress the nerve or the spinal cord causing pain consistent with nerve compression or spinal cord dysfunction, also known as myelopathy.

Lumbosacral radiculopathy is a disorder that causes pain in the lower back and hip which radiates down the back of the thigh into the leg. This damage is caused by compression of the nerve roots which exit the spine at levels of L1- S4. The compression can result in tingling, radiating pain, numbness, paraesthesia, and occasional shooting pain.

A combination of factors including pressure, inflammation, and an immune response seem to be implicated in the pathogenesis of both acute and chronic radicular pain. Pressure would not be a cause of pain, but rather of nerve dysfunction such as weakness and numbness, while the addition of both inflammation and immune response could explain the severe pain experienced by patients suffering from radicular pain.

High power laser therapy (HPLT) is a new, non-invasive, painless, and powerful method with anti-inflammatory and reparative effects. HPLT has therapeutic benefits through photochemical, photothermal, and photomechanical mechanisms, possibly due to its potential for reducing inflammation, enhancing microcirculation, and stimulating immunological proteins and nerve regeneration and secretion of β-endorphins.

MRI: It is the study of choice to visualize herniated disc. MRI findings will help surgeons and other providers plan procedural care if it is indicated. Disc protrusion and nerve root compression can be identified. As Magnetic resonance imaging (MRI) is a medical imaging technique that uses a magnetic field and computer-generated radio waves to create detailed images of the organs and tissues in the body.

Imaging for diagnosis disc herniation are X-rays: These are very accessible at most clinics and outpatient offices. This imaging technique can be used to assess for any structural instability. If x-rays show an acute fracture, it needs to be further investigated using a computed tomogram (CT) scan or magnetic resonance imaging (MRI) .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by orthopedic or neurological consultants depended on MRI assessment as disc herniation (L4-L5/L5-S1levels) with lumbar radiculopathy.
* patients from both genders.
* The patient age will range from 30-45 years old.
* Duration of illness ranged from 3 to 6 months.
* All patients in the study should be ambulant independently.
* Medically and psychologically stable patients.

Exclusion Criteria:

* Previous lumbar or hip surgery.
* Cauda equina syndrome
* Fracture of the bones of lower extremity.
* Major neurological condition (e.g., stroke, multiple sclerosis, Epilepsy, Meningitis, and Brain tumor).
* BMI not more than 30.
* Vascular Impairment.
* Pregnancy and Gynecological problems
* Red flags: spinal tumors, spinal fractures, osteoporosis, infection.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 to 6 months
  Visual Analogue Scale (VAS):
  This scale is used to assess the severity of pain. It consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero) to the worst pain (10) that the patient could feel
Back Pain Related Disability (ODI) using Oswestry low back pain disability questionnaire | 3-6 months
  Modified Oswestry low back disability questionnaire will be used to evaluate patient functional disability. It consists of 10 sections of activities of daily life. Patient asked to answer by checking ONE box in each section for the statement which best applies to her. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5.

CONTACTS AND LOCATIONS:
Overall Officials: ashraf ahmed abdelmonem, md, Study Director — assistant professor of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i will decide later

REFERENCES:
- [Background] Huang Y, Gao D. The effectiveness of high intensity laser therapy in the patients with lumbar disc herniation: A protocol of randomized placebo-controlled trial. Medicine (Baltimore). 2020 Oct 9;99(41):e22520. doi: 10.1097/MD.0000000000022520. PMID 33031293